CLINICAL TRIAL: NCT03337503
Title: Safety and Efficacy of Medical Cannabis Oil in the Treatment of Patients with Chronic Pain: a Randomized, Double-Blind, Placebo-Controlled Pilot Study, Followed by an Open-Label Extension Phase
Brief Title: Safety and Efficacy of Medical Cannabis Oil in the Treatment of Patients with Chronic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to stop the study
Sponsor: Santé Cannabis (Other)
Collaborators: Tetra Bio-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cannabis Oil Study PPP005-001
Record Dates: First submitted 2017-10-17; First posted 2017-11-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- THC and CDB in a 1 to 1 ratio (Experimental): Post a self-titrating schedule of medical cannabis oil, subjects take 1 capsule three times a day at 6 hour intervals.
  2.5 mg THC with 2.5 mg CBD capsule
  Interventions: Drug: THC and CDB in a 1 to 1 ratio
- THC and CBD in a 1 to 2 ratio (Experimental): Post a self-titrating schedule of medical cannabis oil, subjects take 1 capsule three times a day at 6 hour intervals.
  2.5 mg THC with 5 mg CBD capsule
  Interventions: Drug: Experimental: THC and CBD in a 1 to 2 ratio
- high CBD with trace THC (Experimental): Post a self-titrating schedule of medical cannabis oil, subjects take 1 capsule three times a day at 6 hour intervals.
  20 mg CBD with traces of THC
  Interventions: Drug: High CBD with trace THC oil
- placebo (Placebo Comparator): Post a self-titrating schedule of carrier oil, subjects take 1 capsule three times a day at 6 hour intervals.
  carrier oil capsule
  Interventions: Other: placebo

INTERVENTIONS:
Drug: THC and CDB in a 1 to 1 ratio — capsule containing cannabis oil
  Arms: THC and CDB in a 1 to 1 ratio
Drug: Experimental: THC and CBD in a 1 to 2 ratio — capsule containing cannabis oil
  Arms: THC and CBD in a 1 to 2 ratio
Drug: High CBD with trace THC oil — capsule containing cannabis oil
  Arms: high CBD with trace THC
Other: placebo — carrier oil capsule
  Arms: placebo

SUMMARY:
Seeking for effective therapeutic strategies, the investigators are proposing to test the effectiveness of different formulations of medical cannabis oil to alleviate chronic pain, which was partially relieved with conventional prescriptions. Furthermore, the investigators would like to assess the effect of different formulations of medical cannabis oil on other symptoms associated to chronic pain like anxiety and depression, as well as insomnia and appetite. Finally, as recently recommended for clinical studies on medical cannabis, the investigators will examine the safety profile of different cannabis formulations focusing on the following elements: a real chronic administration with more than two weeks of treatment, a larger number of patients, and the clinical relevance of medical cannabis oil to change the amount and type of concomitant medications used to control chronic non-cancer and cancer pain.

DETAILED DESCRIPTION:
This is a 6-week randomized, double-blind, placebo-controlled, parallel group design trial followed by an open-label extension phase of 12 weeks, to evaluate the safety and efficacy of different formulations of medical cannabis oil to reduce chronic pain intensity.

The study will be conducted at Santé Cannabis Clinic, the only medical cannabinoid therapy clinic, located in Montreal, Quebec. One hundred and sixty consecutive adult patients, male and female, with chronic non-cancer and cancer pain (at least 3 months in duration), with an average weekly pain intensity score greater than 4 on the 11 points NRS, will be prospectively recruited and invited to participate in this trial.

Informed consent will be obtained by a Research Assistant.

After baseline documentation with standardized scales, patients will be randomized to one of 4 parallel groups:

* Group A: THC/CBD ratio 1:1 capsule
* Group B: THC/CBD ratio 1:2 capsule
* Group C: THC/CBD ratio 0.1:2 capsule
* Group D: Placebo capsule Patients will have a dose titration phase during the first week. The dose escalation will allow patients to adapt to the potential adverse effects (AEs) of the medical cannabis.

Follow-up visits will be done after 1 week and 6 weeks of treatment. At the end of the first phase of the study, patients who wish to participate in the open-label extension phase will have the option to continue in the same treatment regimen. For the placebo group, the investigator may propose one of the cannabis oils to the subject if they feel it may potentially provide benefits.

They will take this new treatment for other 12 weeks. For this open-label extension phase the follow-up visits will be done after 4 weeks and 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Adult patients (older than 18 years of age), male and female, with chronic non-cancer and cancer pain (at least 3 months in duration)
3. Patients experiencing an average weekly pain intensity score greater than 4 on a 11 points NRS
4. Subject agreed to follow the protocol
5. Naïve cannabis patients with chronic non-cancer and cancer pain (not used cannabis in any presentation in the last 12 weeks)
6. Patients receiving opioids and other concomitant pain medications should have a stable dose for the last 15 days.
7. Normal cognitive status according to MiniCog
8. Normal liver function (defined as aspartate aminotransferase 10-40 U/L and alanine aminotransferase 7-56 U/L)
9. Normal renal function (defined as serum creatinine level <133 µmol/L and Estimated Glomerular Filtration Rate (eGFR) greater than or equal to 60)
10. Negative result on βhuman chorionic gonadotropin pregnancy test (if applicable)
11. Ability to read and respond to questions in French or English.
12. A female volunteer must meet one of the following criteria:

    If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first drug administration, during the study and for at least 60 days after the last dose.

    If of non-childbearing potential - should be surgically sterile or in a menopausal state
13. A male volunteer with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must be surgically sterile or agrees to use one of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration.

Exclusion Criteria:

1. Acute pain (less than 3 months in duration)
2. Previous serious adverse event or hypersensitivity to cannabis or cannabinoids
3. Inability to understand and comply with the instructions of the study
4. Presence of significant cardiac disease (history of unstable ischemic heart disease, heart failure, severe and uncontrolled hypertension) that, in the opinion of the investigator, would put the patient at risk of a clinically significant arrhythmia or myocardial infarction
5. Current substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM 5)
6. Life-time history of dependence on cannabis or diagnosis of cannabis use disorder (CUD) according to the DSM 5
7. Life-time history of DSM 5 schizophrenia, bipolar disorder, or previous psychosis with or intolerance to cannabinoids
8. Current or history of suicidal ideation
9. Pregnant, breast-feeding or female patients of child-bearing potential and male patients whose partner is of child-bearing potential, unless willing to ensure that they or their partner use effective contraception
10. Hepatic impairment (aspartate aminotransferase more than three times normal) or renal function impairment (serum creatinine level >133 µmol/L, Estimated Glomerular Filtration Rate (eGFR) <60)
11. Cognitive impairment according to MiniCog
12. The patient is currently using or has used cannabinoid based medications within 90 days of study entry and is unwilling to abstain for the duration of the study
13. Positive urine drug screen for cannabinoids and other potential abuse substances (e.g. alcohol, cocaine, amphetamines and methamphetamines, unprescribed opioids)
14. Participation in another clinical trial within 30 days of enrolment in our trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Does the daily use of cannabis oil improves chronic pain | Change from Baseline in BPI-SF at Weeks 1 and 6 and in follow-up phase at Weeks 10 and 18.
  Changes in pain as measured by the Brief Pain Inventory-Short Form (BPI-SF) scale. Scale range is 0 to 10; 0 (No pain) being the best rating to the maximal rating of 10 (Pain as bad as you can imagine).
Does the daily use of cannabis oil improves chronic pain | Change from Baseline in NRS at Weeks 1 and 6 and in follow-up phase at Weeks 10 and 18.
  Changes in pain as measured by the Numerical Rating Scale (NRS). The NRS is a measure of the average weekly pain intensity score greater than on a 0 to 10 points scale where 0 is No Pain and 10 is the worst pain.

SECONDARY OUTCOMES:
Does the daily use of cannabis oil improve symptom burden | Change from Baseline in ESAS-r-CS at Weeks 1 and 6 and in follow-up phase at Weeks 10 and 18.
  Changes in symptom burden as measured by the revised Edmonton Symptom Assessment System version with Constipation and Sleep was added to assess improvement in symptom burden (ESAS-r-CS). Scale range is 0 to 10; 0 (No symptom) being the best rating to the maximal rating of 10 (Worst possible score for symptom).
Does the daily use of cannabis oil reduce the severity of Treatment-Emergent Adverse Events (safety and tolerability). | Change from Baseline in UKU-SERSP at Weeks 1 and 6 and in follow-up phase at Weeks 10 and 18.
  Changes in validated UKU Side Effects Rating Scale for Patients (UKU-SERS-Pat). Scale range is 0 to 3 for rating the degree of severity and a second scale for the investigator that assigns a casual relationship of improbable, possible or probable.
Does the daily use of cannabis oil improve cognition | Change from Baseline in Mini-Cog at Weeks 1 and 6 and in follow-up phase at Weeks 10 and 18.
  Changes in validated Mini-Cog. Scale range is numerical and rates the ability to recall words and ability to draw a clock showing numbers from 1 to 12 and then drawing the given time.
Does the daily use of cannabis oil reduce the Profile of Mood States (POMS) | Change from Baseline in POMS at Weeks 1 and 6 and in follow-up phase at Weeks 10 and 18.
  Changes in POMS . Scale range is 1 to 5 and describes how you feel right now. Scale of 1, the lowest score, describes a feeling of Not At All right now for the mood and the scale of 5 gives the highest score representing a feeling of Extremely for the mood.
Does the daily use of cannabis oil improve the Hamilton Rating Scale for Depression (HAM-D) | Change from Baseline in HAM-D at Weeks 1 and 6 and in follow-up phase at Weeks 10 and 18.
  Changes in HAM-D scale. Scale range is either 0 to 2 or 0 to 4. The scale is designed to rate the severity of depression with a score of 0 representing the absence of the question and 2 or 4 meaning the highest severity.
Does the daily use of cannabis oil improve Medication Quantification Scale (MQS) version III | Change from Baseline in MQS version III at Weeks 1 and 6 and in follow-up phase at Weeks 10 and 18.
  Changes in concurrent medications, rescue medications and Medication Quantification Scale (MQS) version III. MQS is a method of quantifying different pain drug regimens by evaluating the use of 22 distinct drug classes (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs], antidepressants, benzodiazepines, opiates). A single value is calculated based on a patient's pain medication profile, taking into account dosages, and the types of pain medications prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Vigano, MD, MSc, Principal Investigator — McGill University; Maria Fernanda Arboleda, MD, Study Director — McGill University
Locations (1):
- Santé Cannabis, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided